CLINICAL TRIAL: NCT02560792
Title: Tailored Activity Goals - an Exercise Prescription Study
Acronym: TAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: F31MH079636 (NIH); F31MH079636 (NIH)
Record Dates: First submitted 2015-07-30; First posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Physical Activity; Affect
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Positive Affect Condition (Experimental): Participants read that their exercise prescription was a healthy level of intensity for exercise, and then read that most people indicated this level of intensity leads to positive affect. To further encourage participants to think about how the supposed typical affective response might apply to them personally, they were also asked to describe how they thought the exercise might lead to positive feelings.
  Interventions: Behavioral: Positive Affect Condition
- Negative Affect Condition (Experimental): Participants read that their exercise prescription was a healthy level of intensity for exercise, and then read that most people indicated this level of intensity leads to negative affect. To further encourage participants to think about how the supposed typical affective response might apply to them personally, they were also asked to describe how they thought the exercise might lead to negative feelings.
  Interventions: Behavioral: Negative Affect Condition
- Control Condition (Experimental): Participants read that their exercise prescription was a healthy level of intensity for exercise - affect was not mentioned.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Positive Affect Condition — Participants read: "Most people exercising at this intensity say that it feels good, and that it makes them feel energized and more positive, and more relaxed afterwards. Thinking about your exercise prescription, please list the reasons or ways in which you, personally, might expect this exercise to lead to positive feelings, and what specifically about this exercise might make you, personally, feel good."
  Arms: Positive Affect Condition
Behavioral: Negative Affect Condition — Participants read: "Most people exercising at this intensity say that it doesn't feel very good, and that it makes them feel tired and not so positive, and not very relaxed afterwards. Thinking about your exercise prescription, please list the reasons or ways in which you, personally, might expect this exercise to lead to negative feelings, and what specifically about this exercise might make you, personally, feel bad."
  Arms: Negative Affect Condition
Behavioral: Control Condition — Participants receive no information about affective response
  Arms: Control Condition

SUMMARY:
The primary goal of this study is to determine experimentally the relationship between affective response to exercise and future exercise behavior. A secondary goal is to examine potential mediators and moderators of this relationship, specifically four variables considered to contribute to the volitional control of exercise behavior - planning, attention, resource commitment, and affect regulation. An additional goal is to examine how symptoms of depression might influence the affective response to exercise, and the relationship between affective response to exercise and exercise behavior.

DETAILED DESCRIPTION:
The specific aims are as follows:

Aim 1. The first aim is to determine the effectiveness of an experimental manipulation of individuals' affective response to a laboratory-supervised bout of exercise corresponding to a vigorous intensity (just below the ventilatory threshold), compared to a control condition that simply measures individuals' natural affective response to exercise. The investigators will specifically determine the effect of this manipulation on anticipated, experienced and remembered affective response to exercise.

Aim 2. The second aim is to examine individuals' adherence to an exercise prescription over the course of one week that asks them to exercise daily on their own for twenty minutes at the same intensity (as indicated by a heart rate monitor) as the laboratory-supervised exercise session, and to determine whether adherence to this prescription is greater for those who expect exercise to lead to positive affect than those who expect exercise to lead to negative affect, as compared to a control condition.

Aim 3. The third aim is to examine potential mediators and moderators of the relationship between anticipated affect and subsequent exercise behavior, including volitional control of exercise, affect regulation ability, and symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* eligible participants will be between the ages of 18 and 39 (for men) and 18 and 45 (for women)
* free of overt disease (as cleared by clinical translational research center medical staff)
* free of mental health conditions other than depression and anxiety (by self-report)
* physically capable of engaging in moderate exercise activity (i.e., no injuries or physical impairments)
* willing to receive a "prescription" for exercise intensity, frequency, and duration, and have access to a computer with Internet connectivity in order to complete the online follow-up survey.

Exclusion Criteria:

* elite (i.e., paid) athletes or required to participate in aerobic exercise in conjunction with their occupation (e.g., aerobics instructors)
* women must not be pregnant or planning to become pregnant during the study period
* on any medications for which exercise is contraindicated (as cleared by clinical translational research center medical staff)
* smoker

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Days of exercise according to prescription as measured by exercise log | 7 days
  Number of days of prescribed exercise recorded on exercise log
Days of exercise according to prescription as measured by heart rate monitor | 7 days
  Number of days of prescribed exercise recorded by heart rate monitor

SECONDARY OUTCOMES:
Intentions to exercise according to prescription as measured by intention to exercise scale | 5 minutes post-intervention
  Self-report survey: intention to exercise scale
Volitional control of exercise: Planning as measured by exercise planning scale | 7 days post-intervention
  Self-report survey: exercise planning scale
Volitional control of exercise: Commitment as measured by commitment to exercise scale | 7 days post-intervention
  Self-report survey: commitment to exercise scale

OTHER OUTCOMES:
Positive activated affect as measured by Physical Activity Affect Scale | 5 minutes before, 10 and 20 minutes during, and 5 minutes after intervention
  Self-report survey: Physical Activity Affect Scale, positive affect subscale
Negative activated affect as measured by Physical Activity Affect Scale | 5 minutes before, 10 and 20 minutes during, and 5 minutes after intervention
  Self-report survey: Physical Activity Affect Scale, negative affect subscale
Tranquility as measured by Physical Activity Affect Scale | 5 minutes before, 10 and 20 minutes during, and 5 minutes after intervention
  Self-report survey: Physical Activity Affect Scale, tranquility subscale
Fatigue as measured by Physical Activity Affect Scale | 5 minutes before, 10 and 20 minutes during, and 5 minutes after intervention
  Self-report survey: Physical Activity Affect Scale, fatigue subscale

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Kwan, PhD, Principal Investigator — University of Colorado School of Medicine